CLINICAL TRIAL: NCT03437161
Title: A Prospective Trial to Compare Deep Inspiratory Breath Hold (DIBH) With Prone Breast Irradiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-01477; s16-01477 (Other: New York University School of Medicine)
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Radiation; Prone position; Supine position; DIBH; Invasive Breast Carcinoma; Ductal Breast Carcinoma In Situ
MeSH Terms: conditions — Breast Neoplasms; Deception; Carcinoma, Intraductal, Noninfiltrating | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation Therapy (RT) (Experimental): Patients attend a simulation visit and undergo two CT scans, one in the prone position and one in the supine position with DIBH. Within 1 week after the simulation visit, patients undergo radiation therapy either in the supine position with DIBH or in the prone position daily for 15-30 consecutive days as per physician's prescription.
  Interventions: Radiation: Radiation Therapy (RT)

INTERVENTIONS:
Radiation: Radiation Therapy (RT) — Undergo RT either in the supine position with DIBH or in the prone position.
  Other Names: Cancer Radiotherapy; Radiotherapy; RT

SUMMARY:
This phase II trial studies how well deep inspiratory breath hold or prone breast radiation therapy works in reducing cardiac dose in patients with breast cancer or ductal carcinoma in situ. Deep inspiratory breath hold is a technique that involves a patient holding their breath during radiation to move the heart away from the breast to minimize radiation to the heart. Prone breast radiation therapy is a technique in which a patient receives treatment "face-down" to minimize the radiation to the rest of the body, including the heart and lungs. Comparing deep inspiratory breath hold to prone breast radiation therapy may help doctors improve radiation to the target while reducing radiation to healthy tissues surrounding the target.

DETAILED DESCRIPTION:
Patients attend a simulation visit and undergo two CT scans, one in the prone position and one in the supine position with DIBH. Within 1 week after the simulation visit, patients undergo radiation therapy either in the supine position with DIBH or in the prone position daily for 15-30 consecutive days as per physician's prescription

ELIGIBILITY:
Inclusion Criteria:

* Any woman with biopsy proven left breast DCIS or invasive cancer who has undergone a lumpectomy and who requires whole breast irradiation to the breast alone (and not to any nodal regions) as per the treating radiation oncologist

Exclusion Criteria:

* Previous radiation to the ipsilateral breast
* All pre-menopausal women will require a urine qualitative pregnancy test to exclude pregnancy; pregnant women will be excluded from the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Mean cardiac dose | Up to 6 weeks
  Assess whether the mean cardiac dose in the supine DIBH plan differs from the mean cardiac dose in the prone plan within strata defined by total RT dose.

SECONDARY OUTCOMES:
Volume of heart receiving > 20 gray (Gy) | Up to 6 weeks
  The volume of heart receiving >20Gy in DIBH plan vs. prone plan
Mean left anterior descending artery (LAD) dose in DIBH plan vs. prone plan | Up to 6 weeks
  The mean LAD dose in DIBH plan vs. prone plan
Maximum left anterior descending artery (LAD) dose in DIBH plan vs. prone plan | Up to 6 weeks
  The maximum LAD dose in DIBH plan vs. prone plan
Mean ipsilateral lung dose | Up to 6 weeks
  The mean ipsilateral lung dose in DIBH plan vs. prone plan
Volume of ipsilateral lung receiving > 20Gy | Up to 6 weeks
  The volume of ipsilateral lung receiving >20Gy in DIBH plan vs. prone plan
Volume of the contralateral breast receiving > 5 Gy | Up to 6 weeks
  The volume of the contralateral breast receiving >5Gy in DIBH plan vs. prone plan
Maximum point dose to planning target volume (PTV) breast | Up to 6 weeks
  The maximum point dose to PTV breast in DIBH plan vs. prone plan
Maximum separation | Up to 6 weeks
  The maximum separation in DIBH plan vs. prone plan
Distance from the mid-sternum to the nipple when the patient is in the prone position | Up to 6 weeks
  Distance from the mid-sternum to the nipple when the patient is in the prone position
PTV breast volume as calculated on the prone scan | Up to 6 weeks
  PTV breast volume as calculated on the prone scan
Change in distance between the chest wall and heart (at the most lateral portion of the chest-wall-heart interface) | Up to 6 weeks
  The change in distance between the chest wall and heart (at the most lateral portion of the chestwall-heart interface) between the free breathing scout films and the DIBH scout films
Patient treatment plan (supine with DIBH or prone) | Up to 6 weeks
  Will be described by proportions and frequency distributions. Logistic regression will be used to assess how each of the covariates (primary and secondary endpoints) affects the probability of being selected to undergo RT using the supine DIBH plan. ROC curves will be generated for various cut-points of the true proportion of patients requiring the supine DIBH plan.

CONTACTS AND LOCATIONS:
Overall Officials: Naamit Gerber, MD, Principal Investigator — Laura and Isaac Perlmutter Cancer Center at NYU Langone